CLINICAL TRIAL: NCT03470363
Title: Effect of Spinal or Sevoflurane Anesthesia on Neutrophil Activation After Tourniquet Induced Ischemia-reperfusion in Knee Surgery
Brief Title: Effect of Spinal or Sevoflurane Anesthesia on Neutrophil Activation During Knee Surgery With Pneumatic Tourniquet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Gregory Minguet, Medical Doctor, Anesthesiologist, Principal Investigator, University of Liege
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 456
Record Dates: First submitted 2018-03-12; First posted 2018-03-19 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Knee Surgery With Tourniquet
Keywords: total knee arthroplasty; tourniquet; sevoflurane; spinal anesthesia; myeloperoxidase; elastase; neutrophil
MeSH Terms: interventions — Bupivacaine; Sufentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Spinal anesthesia (Active Comparator): Knee surgery under spinal anesthesia
  Intervention involves spinal administration of 12,5 mg bupivacaine and 2,5 microgram sufentanil.
  Interventions: Drug: Bupivacaine / SUFentanil
- Group Sevoflurane anesthesia (Active Comparator): Knee surgery under sevoflurane anesthesia
  Intervention involves administration of inhaled sevoflurane for maintenance of general anesthesia
  Interventions: Drug: Sevoflurane Volatile Liquid

INTERVENTIONS:
Drug: Sevoflurane Volatile Liquid
  Arms: Group Sevoflurane anesthesia
Drug: Bupivacaine / SUFentanil
  Arms: Group Spinal anesthesia

SUMMARY:
Aim of study : Assessement of neutrophil activation during ischemia reperfusion associated with tourniquet use for total knee arthroplasty. This activation was compared in a group of patient scheduled for spinal anesthesia and for sevoflurane anesthesia

DETAILED DESCRIPTION:
Aim of study : Assessement of neutrophil activation during ischemia reperfusion associated with tourniquet use for total knee arthroplasty. This activation was compared in a group of patient scheduled for spinal anesthesia and for sevoflurane anesthesia This activation was assessed by plasma myeloperoxidase and elastase measurements in four consecutive blood samples during and after surgery (before surgical incision and 1, 3, 24 hours following tourniquet release.

ELIGIBILITY:
Inclusion Criteria:

* Total knee arthroplasty under spinal or sevoflurane anesthesia

Exclusion Criteria:

* American Society of Anesthesiologists class 3 and 4
* vascular disease of the lower limbs
* cardiac or respiratory disease
* immune disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Changes in plasmatic concentration of myeloperoxidase and elastase | Before surgical incision and one hour after tourniquet release
  Biological measurement of changes in plasmatic concentration of myeloperoxidase and elastase from preoperative values to one hour after tourniquet release.
Changes in plasmatic concentration of myeloperoxidase and elastase | Before surgical incision then 3 and 24 hours after tourniquet release
  Biological measurement of changes in plasmatic concentration of myeloperoxidase and elastase from preoperative values to 3 and 24 hours after tourniquet release.

SECONDARY OUTCOMES:
Changes in plasmatic concentration of endothelial biomarkers | Before surgical incision and one hour after tourniquet release
  Biological measurement of changes in plasmatic concentration of syndecan-1, soluble thrombomodulin, soluble E-selectin and VEGF from preoperative values to one hour after tourniquet release.
Changes in plasmatic concentration of endothelial biomarkers | Before surgical incision then 3 and 24 hours after tourniquet release
  Biological measurement of changes in plasmatic concentration of syndecan-1, soluble thrombomodulin, soluble E-selectin and VEGF from preoperative values to 3 and 24 hours after tourniquet release.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Brichant, MD, PhD, Study Chair — University of Liege

IPD SHARING:
Plan to Share IPD: No